CLINICAL TRIAL: NCT01101620
Title: Pilot Study on the Effects of Levosimendan on in Vivo Respiratory Muscle Function in Healthy Subjects
Brief Title: Effect of Levosimendan on Respiratory Muscle Function in Healthy Subjects
Acronym: LSD1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Nijmegen (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Leo Heunks, University Medical Center Nijmegen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Levo1
Record Dates: First submitted 2010-04-09; First posted 2010-04-12 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2010-09

CONDITIONS: Respiratory Muscle Function
MeSH Terms: interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levosimendan (Active Comparator)
  Interventions: Drug: Levosimendan
- Placebo (Placebo Comparator)
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan

SUMMARY:
The purpose of this study is to investigate if levosimendan improves contractile performance of the diaphragm in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* informed consent

Exclusion Criteria:

* use of any prescript medication
* chronic hiccups
* pre-existent muscle disease (congenital or acquired) or diseases / disorders know to be associated with myopathy including diabetes and auto-immune diseases.
* pre-existent lung disease
* pre-existent cardiac disease (based on history, electrocardiography and transthoracic echocardiography)
* pregnancy, breast feeding
* upper airway / esophageal pathology
* phrenic nerve lesions
* any metals in body (pacemaker, splinters, metal stiches)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Contractility of the diaphragm elicited with magnetic stimulation of the phrenic nerves | Multiple measurements within 4 hours after administration of study medication
Fatiguability of the diaphragm | Multiple measurements within 4 hours after administration of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Leo Heunks, MD, Principal Investigator — University Medical Center Nijmegen; Jonne Doorduin, Principal Investigator — University Medical Center Nijmegen
Locations (1):
- University Medical Center Nijmegen, Nijmegen, Gelderland, Netherlands